CLINICAL TRIAL: NCT06821815
Title: The Effect of Intensive Video-Based Game Therapy Applications on Motor Skills, Daily Living Activities and Participation in Cerebral Palsy
Brief Title: Intensive Video-Based Game Therapy Applications in Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ahmet Emir, DR, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7476
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Palsy (CP)
Keywords: video game based therapy; cerebral palsy; bimanual therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Exergaming

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessor of the study protocol wont be able to have knowledge about assigned group of participants.
  Participants wont be aware about groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video Game Based Therapy Group (Experimental): In this group an Intensive video game based therapy program will be applied to participants. Therapy program aimed for the motor function of upper extremities and postural control. Therapy program includes 10 individual 4 group sessions per week, 28 sessions in total with each session lasts 40 minutes. Total duration of this intervention is 2 weeks.
  Interventions: Other: Video Game Based Therapy
- Bimanual Intensive Therapy Group (Active Comparator): In this group an Bimanual Intensive therapy program will be applied to participants. Therapy program aimed for the motor function of upper extremities and postural control. Therapy program includes 10 individual 4 group sessions per week, 28 sessions in total with each session lasts 40 minutes. Total duration of this intervention is 2 weeks.
  Interventions: Other: Bimanual Intensive Therapy

INTERVENTIONS:
Other: Video Game Based Therapy — Video game based therapy interventions includes active video games for rehabilitation. Leap Motion Controller based rehabilitative games, Xbox Kinect Games and Kinect Based Custom Rehabilitative Games will be applied to the participants
  Other Names: Virtual Reality; Active Video Game; Exergame
  Arms: Video Game Based Therapy Group
Other: Bimanual Intensive Therapy — This intervention includes goal directed activity based exercises for upper extremity functions. This intervention also includes exercises for postural control
  Arms: Bimanual Intensive Therapy Group

SUMMARY:
This study investigates the effectiveness of intensive video game-based rehabilitation and intensive bimanual activity-based therapy for improving motor skills and daily living activities in individuals with spastic cerebral palsy (CP). Given the importance of high-frequency, short-duration interventions in CP rehabilitation, the research compares these two approaches while ensuring participants receive no additional therapy during the study.

Twenty children (ages 4-18) with GMFCS levels 1-2 and MACS levels 1-3 will be randomly assigned to one of the two groups. The video game-based group will complete 28 structured sessions over two weeks, including 20 individual sessions and 8 group sessions. The control group will follow an identical schedule using bimanual goal-oriented activities. Assessments will be conducted before, after, and three months post-intervention using validated motor and functional performance measures.

By standardizing task contents between groups, the study aims to provide objective results and contribute to CP rehabilitation by identifying an effective, time-efficient, and cost-effective therapy option using exergames and serious games.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is the most common physical disability observed in childhood. Due to the motor function losses observed in individuals with CP, their participation in activities is restricted. Rehabilitation approaches applied to develop motor skills and functional independence in individuals with CP are currently implemented with a target-oriented approach based on motor learning. In this context, video game-based rehabilitation programs are also frequently applied today. The principles of implementation, therapy durations, and session frequencies of motor learning-based rehabilitation approaches in CP rehabilitation vary in the literature. Most application methods are applied over a long period. However, nowadays, it is important to apply these therapy practices for a shorter duration but with high session frequency and intensity to achieve motor skill and functional independence goals in a shorter time.In light of this information, the study aims to investigate the effectiveness of an intensive video game-based rehabilitation program and an intensive bimanual activity-based therapy program for motor skills and daily living activities in individuals with CP. Applying video game-based rehabilitation programs in an intensive format to achieve the targeted functional improvements in upper extremity functions and motor skills in a short time and comparing the effectiveness of this approach with another intensive therapy program, while ensuring that the groups do not receive any other rehabilitation approach during the application period, makes our study unique. The study will include 20 children diagnosed with spastic cerebral palsy, aged 4-18, with Gross Motor Function Classification System (GMFCS) levels 1-2, Manual Ability Classification System (MACS) levels 1-3, who can follow given visual and verbal commands, Communication Function Classification System (CFCS) levels 1-2, Visual Function Classification System (VFCS) levels 1-2, who continue the program within the specified times, and who agree not to receive any therapy other than the one assigned randomly to their group during the study and sign the consent form. In the study, before, after, and 3 months after the 2-week rehabilitation program, assessments will be made using a demographic form, Gross Motor Function Measure-88 (GMFM-88), Canadian Occupational Performance Measure (COPM), Pediatric Evaluation of Disability Inventory Computer Adaptive Test (PEDI-CAT), Box & Block Test, Upper Extremity Selective Motor Control Scale (SCUES), and Becure Balance System. The study group will receive a total of 28 sessions of intensive and structured video game-based rehabilitation, consisting of 20 individual sessions (5 days a week, 2 sessions per day, each session lasting 30-45 minutes) and 8 group training sessions over 2 weeks. The control group will also follow the same plan for 2 weeks, receiving a total of 28 sessions of intensive bimanual goal-oriented activity-based intervention. Care will be taken to ensure that the task contents applied between the two programs are similar to obtain objective results. The therapeutic approach determined and applied during this project, designed with exergames and serious games, is expected to guide professionals working in the field of CP. In this way, it will be possible to find solutions to patients' problems with the most effective and fastest treatment option and at a lower cost.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Spastic Cerebral Palsy
* Gross Motor Function Classification level I-II
* Manual Ability Classification level I-III
* Communication Function Classification System I-II
* No botox injections 6 months prior to the intervention

Exclusion Criteria:

* Visual problems which may effect the interventions
* Secondary conditions such as intellectual disability, epilepsy
* Having surgical procedure related to musculoskeletal system 1 year prior to he study

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
Gross Motor Function changes over the Study - Gross Motor Performance Measure - 88 (GMFM-88) | Prior to the interventions, right after the 2 weeks of interventions and 2 months later as follow-up
  GMFM-88 is a assessment tool to evaluate gross motor functions in children with cerebral palsy. It evaluates motor functions in 5 dimensions and with 88 items total
Performance of Activities of Daily Living - Canadian Occupational Performance Measure (COPM) | Prior to the interventions, right after the 2 weeks of interventions and 2 months later as follow-up
  The Canadian Occupational Performance Measure (COPM) is a client-centered assessment tool that evaluates self-perceived performance and satisfaction in daily activities across three areas: self-care, productivity, and leisure. Clients identify up to five important but challenging activities and rate their performance and satisfaction on a 10-point scale (1 = extremely poor/not satisfied, 10 = excellent/completely satisfied). The total performance and satisfaction scores are averaged separately, with higher scores indicating better function and greater satisfaction. A change of 2 or more points is considered clinically significant.

SECONDARY OUTCOMES:
Changes on Motor Function for Upper Extremities - Selective Control of the Upper Extremity Scale (SCUES) | Prior to the interventions, right after the 2 weeks of interventions and 2 months later as follow-up
  The Selective Control of the Upper Extremity Scale (SCUES) is a clinical tool used to assess selective motor control in the upper extremities of individuals with neurological impairments, particularly cerebral palsy (CP). It evaluates a person's ability to voluntarily isolate and control specific upper limb movements without involuntary muscle activation. SCUES assesses six movement patterns (shoulder flexion/extension, elbow flexion/extension, forearm supination/pronation, wrist flexion/extension) on a 3-point scale: 0 = no selective control, 1 = partial control, 2 = full selective control. Scores from each movement are summed, with a higher total score indicating better selective motor control. SCUES is useful for tracking motor function changes and evaluating the effectiveness of interventions aimed at improving upper limb movement in individuals with CP.
Changes on Motor Function for Upper Extremities - Box and Block Test | Prior to the interventions, right after the 2 weeks of interventions and 2 months later as follow-up
  The Box and Block Test (BBT) is a standardized assessment used to measure manual dexterity and upper limb function in individuals with neurological impairments, including cerebral palsy (CP). The test involves transferring as many small blocks as possible from one compartment of a box to another in 60 seconds, using one hand at a time. The score is the total number of blocks successfully moved, with higher scores indicating better fine motor coordination, speed, and dexterity. The BBT is widely used in rehabilitation to track motor function progress and evaluate the effectiveness of interventions targeting upper limb performance.

OTHER OUTCOMES:
Change of Postural Control | Prior to the interventions, right after the 2 weeks of interventions and 2 months later as follow-up
  The Becure balance system will be used for the Postural Control Assessment. It is custom made assessment system uses wii balance board. Centre of Gravity (COG) displacement and velocity of COG will be collected datas.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Emir, Emir, Principal Investigator — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Cerebral Palsy Türkiye Foundation, Istanbul, Ataşehir
  - Istanbul Medipol University, Istanbul, Beykoz

IPD SHARING:
Plan to Share IPD: Undecided
We are willing to share data of study, only by requests for meta analysis studies.

REFERENCES:
- [Background] Bleyenheuft Y, Arnould C, Brandao MB, Bleyenheuft C, Gordon AM. Hand and Arm Bimanual Intensive Therapy Including Lower Extremity (HABIT-ILE) in Children With Unilateral Spastic Cerebral Palsy: A Randomized Trial. Neurorehabil Neural Repair. 2015 Aug;29(7):645-57. doi: 10.1177/1545968314562109. Epub 2014 Dec 19. PMID 25527487